CLINICAL TRIAL: NCT05683717
Title: A Phase I, Multicenter, Open Label, and Dose-Escalation Study of TT-01488, Administered Orally in Adult Patients With B-Cell Malignancies
Brief Title: A Phase 1 Study to Evaluate the Safety and Tolerability of TT-01488 in Patients With B-Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TT01488CN02
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: B-Cell Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation for TT-01488 (Experimental): TT-01488 tablets will be administered once daily in a 28-day cycle in increasing strength in order to determine the recommended dose for dose expansion.
  Interventions: Drug: TT-01488 Tablets
- Dose Expansion for TT-01488 (Experimental): TT-01488 tablets will be administered once daily in 28-day cycles to verify the safety and preliminary efficacy as observed in the dose escalation cohorts.
  Interventions: Drug: TT-01488 Tablets

INTERVENTIONS:
Drug: TT-01488 Tablets — TT-01488 tablet will be administered orally once daily per protocol defined schedule.

SUMMARY:
This is a multicenter, open-label Phase I dose escalation study to evaluate the safety and preliminary efficacy of the TT-01488 tablet, a non-covalent reversible BTK inhibitor, for the treatment of adult patients with B-cell malignancies.

DETAILED DESCRIPTION:
The study will consist of two parts, dose escalation and dose expansion. A modified 3+3 design will be used to guide the dose escalation and the determination of the dose recommended for dose expansion (DRDE). A sentinel cohort comprising of one subject will be enrolled at a starting dose of 50 mg q.d. Subsequently, patients will be enrolled according to the standard 3+3 dose escalation design to determine the DRDE. Once the DRDE has been selected, TT-01488 of DRDE will be further tested in the dose expansion cohort to verify the safety and preliminary efficacy as observed in the dose escalation cohorts. A recommended Phase II dose (RP2D) may be determined based on the totality of safety, pharmacokinetics, and efficacy data from the dose escalation cohorts and dose expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed B-cell malignancy, failed or intolerant to either ≥ 2 prior standard/common regimens given in combination or sequentially OR have received 1 prior BTK-containing regimen, relapse/refractory, and with treatment indication:

  * CLL/SLL treated with prior immunochemistry or BTK inhibitor containing regimen;
  * DLBCL treated with prior CD20 or anthracyclines containing regimen;
  * Other types of B-cell NHL treated with prior CD20 containing regimen
* Adequate organ function, defined by the following laboratory parameters:

  * Hematologic:
* Absolute neutrophil count (ANC) ≥ 0.75×10^9/L, and ≥ 0.5×10^9/L if bone marrow involved
* Platelets ≥ 50×10^9/L without transfusion within 7 days, and ≥ 30×10^9/L if bone marrow involved
* Hemoglobin ≥ 8.0 g/dL without transfusion within 7 days, and ≥ 7.0 g/dL if bone marrow involved

  * Coagulation:
* Prothrombin time (PT) ≤ 1.5 × ULN
* Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN

  * Renal function:
* Creatinine clearance ≥ 30 mL/min estimated glomerular filtration rate based on Cockcroft-Gault formula

  * Liver function:
* Total bilirubin ≤ 1.5 × ULN (unless due to Gilbert's disease)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 × ULN unless disease-related

Exclusion Criteria:

* Women who are pregnant or lactating
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease-free for at least 2 years or which will not limit survival to < 2 years (Note: these cases must be discussed with the Medical Monitor and/or Investigator)
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or significant screening ECG abnormalities
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified T-cell (CAR-T) therapy within the past 60 days or with any of the following:

  * Active graft versus host disease (GvHD);
  * Cytopenias from incomplete blood cell count recovery post-transplant;
  * Need for anti-cytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity > Grade 1 from CAR-T therapy;
  * Ongoing immunosuppressive therapy
* Grade ≥ 2 toxicity (other than alopecia) continuing from prior anticancer therapy, including radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) of TT-01488 | Up to 28 days after first dose
  Safety and tolerability of TT-01488 as a single agent
Dose recommend for dose expansion (DRDE) | 3 years
  Safety and tolerability of TT-01488 as a single agent
Maximum Tolerated Dose (MTD), if reached, of TT-01488 | Up to 28 days after first dose
  Safety and tolerability of TT-01488 as a single agent

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) | 3 years
  Safety and tolerability of TT-01488 as a single agent. AEs will be assessed per CTCAE v5.0 or 2018 IWCLL and may include, but is not limited to, clinically abnormal laboratory tests, physical exams, vital signs, electrocardiograms, and ECOG performance status.
Area under the concentration time curve (AUC 0-t) | 3 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Maximum plasma concentration (Cmax) | 3 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Time to Maximum Plasma Concentration (Tmax) | 3 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Half-life (T1/2) | 3 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Mean Residence Time (MRT) | 3 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Apparent volume of distribution associated with the terminal phase (Vz/F) | 3 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Apparent clearance (CL/F) | 3 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Objective Response Rate (ORR) | 3 years
  Preliminary efficacy profile of TT-01488 as a single agent
Disease Control Rate (DCR) | 3 years
  Preliminary efficacy profile of TT-01488 as a single agent
Duration of Response (DOR) | 3 years
  Preliminary efficacy profile of TT-01488 as a single agent
Progression free survival (PFS) | 3 years
  Preliminary efficacy profile of TT-01488 as a single agent
Overall survival (OS) | 3 years
  Preliminary efficacy profile of TT-01488 as a single agent

CONTACTS AND LOCATIONS:
Overall Officials: Li Jianyong, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Xu Wei, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No